CLINICAL TRIAL: NCT03774108
Title: Metformin Administration Effect Over Systemic Inflammation Serum Markers in HIV Positive Prediabetic Patients
Brief Title: Metformin and Systemic Inflammation in HIV
Acronym: Metfo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Moises Ramos Solano, Associate professor, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114/18
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: PreDiabetes; HIV-1-infection
MeSH Terms: conditions — Prediabetic State | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Experimental Arm (Experimental): Metformin 850mg/12 hours, oral, 8 weeks
  Interventions: Drug: Metformin Hydrochloride 850 MG
- Placebo Comparator Arm (Placebo Comparator): Placebo pills/12hours, oral, 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride 850 MG — 8 weeks tratment with oral metformin
  Arms: Metformin Experimental Arm
Other: Placebo — 8 weeks tratment with oral placebo
  Arms: Placebo Comparator Arm

SUMMARY:
The purposes of this study are to find out if: metformin can be combined with anti-HIV drugs to reduce systemic inflammation measured by the determination of cytokines and other series of serum markers. To determine if the concomitant administration of metformin with TARA improves the immune function on the CD4 T cell count and its relation with the CD8 T cells, during the treatment and after its interruption.

To this end, in the present study, patients with prediabetes (who meet the fasting impaired glucose criteria) will be identified and treated with metformin or placebo for 8 weeks, receiving stable TARA and with a CD4 + level> 200 cells / μL.

40 patients from the HIV Unit of the Civil Hospital of Guadalajara "Fray Antonio Alcalde" will be included in this study and the intervention will last 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes,
* Age ≥18 years of age
* With a diagnosis of HIV-1 infection,
* That they are receiving TARE for at least 12 months (time necessary to establish a stable reservoir),
* Patients with undetectable viral load (<40 copies / mL) for at least 12 months,
* Have a CD4 + level> 200 cells / μL,
* That they do not have a diagnosis of co-infection with HCV or HBV,
* Patients who do not have a severe alcohol intake (<21 glasses / week in men and <14 glasses / week in women),
* Patients who do not use drugs during the last 90 days prior to the screening visit, or during the study,
* Who wish to participate voluntarily in the study and give their written consent.

Exclusion Criteria:

* Individuals with a known hypersensitivity / allergy to metformin.
* Patients with contraindications to the use of metformin *.
* Individuals who are actively involved in an experimental therapy study or who have received experimental therapy in the last 6 months.
* People suffering from stage IV-V chronic kidney disease, uncontrolled heart failure or active infections.
* Individuals with diabetes mellitus (according to the criteria of the American Diabetes Association *).
* Patients with indication for the use of statins, aspirin or immunomodulators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-01-08 (Estimated)

PRIMARY OUTCOMES:
Quantification of proinflammatory cytokines serum levels by Cytometric Bead Array in prediabetic HIV positive patients after 8 weeks treatment with Metformin | Basal - 8 weeks
  Serum levels of proinflammatory cytokines will be quantify by flow cytometry using a Cytometric Bead Array. The cytokine panel to be messured will be as follows:
  * IL-1beta
  * IFN-alpha2
  * IFN-gamma
  * TNF-alpha
  * MCP-1
  * IL-6
  * IL-8
  * IL-10
  * IL-12p70
  * IL-17A
  * IL-18
  * IL-23
  * IL-33
  These cytokines will be quantify in prediabetic HIV positive patients after 8 weeks treatment with Metformin

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data from participants will be available upon reasonable request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Basal - 8 weeks

REFERENCES:
- [Background] Slim J, Saling CF. A Review of Management of Inflammation in the HIV Population. Biomed Res Int. 2016;2016:3420638. doi: 10.1155/2016/3420638. Epub 2016 Sep 27. PMID 27766258
- [Background] Arafath S, Campbell T, Yusuff J, Sharma R. Prevalence of and Risk Factors for Prediabetes in Patients Infected With HIV. Diabetes Spectr. 2018 May;31(2):139-143. doi: 10.2337/ds17-0009. PMID 29773933
- [Background] Nou E, Lo J, Grinspoon SK. Inflammation, immune activation, and cardiovascular disease in HIV. AIDS. 2016 Jun 19;30(10):1495-509. doi: 10.1097/QAD.0000000000001109. PMID 27058351
- [Background] Saisho Y. Metformin and Inflammation: Its Potential Beyond Glucose-lowering Effect. Endocr Metab Immune Disord Drug Targets. 2015;15(3):196-205. doi: 10.2174/1871530315666150316124019. PMID 25772174